CLINICAL TRIAL: NCT03954158
Title: A Phase 2b, Multi Center, Randomized, Double-Blind, Vehicle-Controlled, Intra-Participant Study, to Evaluate Efficacy and Safety of Two Regimens of Crisaborole Ointment 2% in Japanese Pediatric and Adult Participants (2 Years and Older) With Mild to Moderate Atopic Dermatitis
Brief Title: Study to Assess Efficacy and Safety of Two Regimens of Crisaborole Ointment 2% in Japanese Participants Aged ≥2 Years With Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C3291028
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Results first posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crisaborole ointment 2% once daily (QD) vs vehicle QD (Experimental): intra-participant comparison, treatment will be randomly assigned to target lesion 1 and lesion 2.
  Interventions: Drug: Crisaborole ointment 2%; Drug: Vehicle
- Crisaborole ointment 2% twice daily (BID) vs vehicle BID (Experimental): Intra-participant comparison, treatment will be randomly assigned to target lesion 1 and lesion 2.
  Interventions: Drug: Crisaborole ointment 2%; Drug: Vehicle

INTERVENTIONS:
Drug: Crisaborole ointment 2% — BID regimen
  Arms: Crisaborole ointment 2% twice daily (BID) vs vehicle BID
Drug: Vehicle — BID regimen
  Arms: Crisaborole ointment 2% twice daily (BID) vs vehicle BID
Drug: Crisaborole ointment 2% — QD regimen
  Arms: Crisaborole ointment 2% once daily (QD) vs vehicle QD
Drug: Vehicle — QD regimen
  Arms: Crisaborole ointment 2% once daily (QD) vs vehicle QD

SUMMARY:
This is a Phase 2b, multi-center, randomized, double-blind, vehicle-controlled, intraparticipant study to evaluate efficacy and safety of two regimens of crisaborole ointment 2% in Japanese pediatric and adult participants (cohort 1: 12 years and older, cohort 2: 2 to under 12 years old) with mild to moderate Atopic Dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ages; Cohort 1: 12 years and older at the time of consent. Cohort 2: 2 years to under 12 years old at the time of consent.
* Has confrimed clinical diagnosis of active AD according to Hanifin and Rajka criteria and has at least 6 months history prior to screening and has been clinically stable for more than 1 month
* Has at least 1% and no more than 30% BSA at baseline/Day1, excluding scalp, genitals and groin area
* Has a Investigator's static global assessment (ISGA) score of Mild (2) or Moderate (3) on Day 1.

Exclusion Criteria:

* Has other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Participants had previous treatment with any topical or systemic PDE-4 inhibitor.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Japan (3):
  - Medical Corporation Heishinkai OPHAC Hospital, Osaka, Osaka
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - Sekino Hospital, Toshima-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3291028

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Crisaborole 2% QD + Vehicle QD, Age Group >=12 Years: Participants in this reporting arm were of age greater than or equal to (>=) 12 years. Investigator determined 2 target lesions of same atopic dermatitis (AD) severity in each participant at baseline (Day 1). Crisaborole ointment 2 percent (%) was applied once daily (QD) to 1 of the target lesions and vehicle was applied QD to another target lesion (intra-participant) for 15 days and participants were followed up to maximum of 35 days after the end of treatment (maximum up to Day 50).
- Cohort 1:Crisaborole 2% BID + Vehicle BID,Age Group >=12 Years: Participants in this reporting arm were of age >=12 years. Investigator determined 2 target lesions of same AD severity in each participant at baseline (Day 1). Crisaborole ointment 2% was applied twice daily (BID) to 1 of the target lesions and vehicle was applied BID to another target lesion (intra-participant) for 15 days and participants were followed up to maximum of 35 days after the end of treatment (maximum up to Day 50).
- Cohort 2:Crisaborole 2% QD + Vehicle QD, Age Group 2-11 Years: Participants in this reporting arm were of age 2 to 11 years. Investigator determined 2 target lesions of same AD severity in each participant at baseline (Day 1). Crisaborole ointment 2% was applied QD to 1 of the target lesions and vehicle was applied QD to another target lesion (intra-participant) for 15 days and participants were followed up to maximum of 35 days after the end of treatment (maximum up to Day 50).
- Cohort 2:Crisaborole 2% BID + Vehicle BID,Age Group 2-11 Years: Participants in this reporting arm were of age 2 to 11 years. Investigator determined 2 target lesions of same AD severity in each participant at baseline (Day 1). Crisaborole ointment 2% was applied BID to 1 of the target lesions and vehicle was applied BID to another target lesion (intra-participant) for 15 days and participants were followed up to maximum of 35 days after the end of treatment (maximum up to Day 50).
Period: Overall Study
Arm/Group | Cohort 1: Crisaborole 2% QD + Vehicle QD, Age Group >=12 Years | Cohort 1:Crisaborole 2% BID + Vehicle BID,Age Group >=12 Years | Cohort 2:Crisaborole 2% QD + Vehicle QD, Age Group 2-11 Years | Cohort 2:Crisaborole 2% BID + Vehicle BID,Age Group 2-11 Years
Started | 20 | 21 | 20 | 20
Completed | 20 | 21 | 20 | 20
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were randomized and received >=1 dose of investigational product.
Groups:
- Cohort 1: Crisaborole 2% QD + Vehicle QD, Age Group >=12 Years: Participants in this reporting arm were of age >=12 years. Investigator determined 2 target lesions of same AD severity in each participant at baseline (Day 1). Crisaborole ointment 2% was applied QD to 1 of the target lesions and vehicle was applied QD to another target lesion (intra-participant) for 15 days and participants were followed up to maximum of 35 days after the end of treatment (maximum up to Day 50).
- Cohort 1:Crisaborole 2% BID + Vehicle BID,Age Group >=12 Years: Participants in this reporting arm were of age >=12 years. Investigator determined 2 target lesions of same AD severity in each participant at baseline (Day 1). Crisaborole ointment 2% was applied BID to 1 of the target lesions and vehicle was applied BID to another target lesion (intra-participant) for 15 days and participants were followed up to maximum of 35 days after the end of treatment (maximum up to Day 50).
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Crisaborole 2% QD + Vehicle QD, Age Group >=12 Years | Cohort 1:Crisaborole 2% BID + Vehicle BID,Age Group >=12 Years | Cohort 2:Crisaborole 2% QD + Vehicle QD, Age Group 2-11 Years | Cohort 2:Crisaborole 2% BID + Vehicle BID,Age Group 2-11 Years | Total
Number analyzed (Participants) | 20 | 21 | 20 | 20 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 20 | 20 | 41
  Between 18 and 65 years | 19 | 21 | 0 | 0 | 40
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 17 | 8 | 11 | 47
  Male | 9 | 4 | 12 | 9 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 21 | 20 | 20 | 81
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 20 | 21 | 20 | 20 | 81
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Sign Score (TSS) in Target Lesions at Day 15: Crisaborole Ointment 2% Versus Vehicle
Description: Lesion TSS was an assessment of the target lesion severity, which was based on severity of 4 clinical signs erythema, induration/papulation, excoriation and lichenification. All of these 4 signs were rated on a scale of 0 to 3 (0= none, 1= mild, 2= moderate, 3= severe). These ratings were added to create a total TSS score; ranging from 0 (none) to 12 (most severe), with higher score representing greater severity.
Time Frame: Baseline, Day 15
Population: FAS included all participants who were randomized and received greater than or equal to 1 dose of investigational product.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Crisaborole 2% QD: Age Group >=12 Years: Participants in this reporting arm were of age >=12 years. Investigator determined 2 target lesions of same atopic dermatitis severity in each participant at baseline (Day 1). Crisaborole ointment 2% was applied QD to 1 of the target lesions for 15 days and participants were followed up to 35 days after the end of treatment (maximum up to Day 50).
- Vehicle QD: Age Group >=12 Years: Participants in this reporting arm were of age >=12 years. Investigator determined 2 target lesions of same atopic dermatitis severity in each participant at baseline (Day 1). Vehicle was applied QD to 1 of the target lesions for 15 days and participants were followed up to 35 days after the end of treatment (maximum up to Day 50).
- Crisaborole 2% BID: Age Group >=12 Years: Participants in this reporting arm were of age >=12 years. Investigator determined 2 target lesions of same atopic dermatitis severity in each participant at baseline (Day 1). Crisaborole ointment 2% was applied BID to 1 of the target lesions for 15 days and participants were followed up to 35 days after the end of treatment (maximum up to Day 50).
- Vehicle BID: Age Group >=12 Years: Participants in this reporting arm were of age >=12 years. Investigator determined 2 target lesions of same atopic dermatitis severity in each participant at baseline (Day 1). Vehicle was applied BID to 1 of the target lesions for 15 days and participants were followed up to 35 days after the end of treatment (maximum up to Day 50).
- Crisaborole 2% QD: Age Group 2 to 11 Years: Participants in this reporting arm were of age 2 to 11. Investigator determined 2 target lesions of same atopic dermatitis severity in each participant at baseline (Day 1). Crisaborole ointment 2% was applied QD to 1 of the target lesions for 15 days and participants were followed up to 35 days after the end of treatment (maximum up to Day 50).
- Vehicle QD: Age Group 2 to 11 Years: Participants in this reporting arm were of age 2 to 11. Investigator determined 2 target lesions of same atopic dermatitis severity in each participant at baseline (Day 1). Vehicle was applied QD to 1 of the target lesions for 15 days and participants were followed up to 35 days after the end of treatment (maximum up to Day 50).
- Crisaborole 2% BID: Age Group 2 to 11 Years: Participants in this reporting arm were of age 2 to 11. Investigator determined 2 target lesions of same atopic dermatitis severity in each participant at baseline (Day 1). Crisaborole ointment 2% was applied BID to 1 of the target lesions for 15 days and participants were followed up to 35 days after the end of treatment (maximum up to Day 50).
- Vehicle BID: Age Group 2 to 11 Years: Participants in this reporting arm were of age 2 to 11. Investigator determined 2 target lesions of same atopic dermatitis severity in each participant at baseline (Day 1). Vehicle was applied BID to 1 of the target lesions for 15 days and participants were followed up to 35 days after the end of treatment (maximum up to Day 50).
Arm/Group | Crisaborole 2% QD: Age Group >=12 Years | Vehicle QD: Age Group >=12 Years | Crisaborole 2% BID: Age Group >=12 Years | Vehicle BID: Age Group >=12 Years | Crisaborole 2% QD: Age Group 2 to 11 Years | Vehicle QD: Age Group 2 to 11 Years | Crisaborole 2% BID: Age Group 2 to 11 Years | Vehicle BID: Age Group 2 to 11 Years
Number analyzed (Participants) | 20 | 20 | 21 | 21 | 20 | 20 | 20 | 20
units on a scale
  Baseline | 7.7 (0.36) | 7.5 (0.45) | 7.1 (0.46) | 7.4 (0.48) | 6.2 (0.38) | 6.5 (0.37) | 7.1 (0.45) | 7.3 (0.44)
  Change at Day 15 | -4.5 (0.60) | -2.9 (0.51) | -4.8 (0.53) | -2.7 (0.47) | -3.5 (0.47) | -2.0 (0.50) | -4.7 (0.50) | -2.6 (0.54)
Statistical Analysis 1: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Vehicle QD: Age Group >=12 Years; Change at Day 15, Intra-participant: Mixed effect Model for Repeated Measures (MMRM) included the fixed effect of visit, and the covariance structure UN was used; Test type: Superiority; p = 0.0071, Mixed Models Analysis; Least squares mean of difference = -1.6, 95% CI 2-sided [-2.7 to -0.5], Standard Error of Mean 0.53
Statistical Analysis 2: Comparison: Crisaborole 2% BID: Age Group >=12 Years vs Vehicle BID: Age Group >=12 Years; Change at Day 15, Intra-participant: Mixed effect Model for Repeated Measures included the fixed effect of visit, and the covariance structure UN was used; Test type: Superiority; p = 0.0029, Mixed Models Analysis; Least squares mean of difference = -2.0, 95% CI 2-sided [-3.3 to -0.8], Standard Error of Mean 0.60
Statistical Analysis 3: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Vehicle QD: Age Group 2 to 11 Years; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0250, Mixed Models Analysis; Least squares mean of difference = -1.5, 95% CI 2-sided [-2.7 to -0.2], Standard Error of Mean 0.60
Statistical Analysis 4: Comparison: Crisaborole 2% BID: Age Group 2 to 11 Years vs Vehicle BID: Age Group 2 to 11 Years; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0014, Mixed Models Analysis; Least squares mean of difference = -2.1, 95% CI 2-sided [-3.3 to -0.9], Standard Error of Mean 0.56

2. Secondary Outcome: Change From Baseline in Total Sign Score in Target Lesions at Day 15: Crisaborole Ointment 2% BID Versus Crisaborole Ointment 2% QD
Description: as for outcome 1
Time Frame: Baseline, Day 15
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Crisaborole 2% QD: Age Group >=12 Years | Crisaborole 2% BID: Age Group >=12 Years | Crisaborole 2% QD: Age Group 2 to 11 Years | Crisaborole 2% BID: Age Group 2 to 11 Years
Number analyzed (Participants) | 20 | 21 | 20 | 20
units on a scale | -4.3 [-5.4 to -3.3] | -4.9 [-5.9 to -3.9] | -3.7 [-4.5 to -2.8] | -4.5 [-5.4 to -3.6]
Statistical Analysis 1: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Crisaborole 2% BID: Age Group >=12 Years; Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen, visit, dosing regimen-by-visit interaction, and baseline value and the covariance structure UN was used; Test type: Other; Difference of least squares mean = -0.6, 95% CI 2-sided [-2.0 to 0.9], Standard Error of Mean 0.4295
Statistical Analysis 2: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Crisaborole 2% BID: Age Group 2 to 11 Years; [analysis description as in outcome 2, analysis 1]; Test type: Other; Difference of least squares mean = -0.8, 95% CI 2-sided [-2.1 to 0.4], Standard Error of Mean 0.61

3. Secondary Outcome: Change From Baseline in Total Sign Score in Target Lesions at Day 8: Crisaborole Ointment 2% Versus Vehicle
Description: as for outcome 1
Time Frame: Baseline, Day 8
Population: FAS included all participants who were randomized and received greater than or equal to 1 dose of investigational product. Here, "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Crisaborole 2% QD: Age Group >=12 Years | Vehicle QD: Age Group >=12 Years | Crisaborole 2% BID: Age Group >=12 Years | Vehicle BID: Age Group >=12 Years | Crisaborole 2% QD: Age Group 2 to 11 Years | Vehicle QD: Age Group 2 to 11 Years | Crisaborole 2% BID: Age Group 2 to 11 Years | Vehicle BID: Age Group 2 to 11 Years
Number analyzed (Participants) | 20 | 20 | 21 | 21 | 20 | 20 | 20 | 20
units on a scale
  Baseline | 7.7 (0.36) | 7.5 (0.45) | 7.1 (0.46) | 7.4 (0.48) | 6.2 (0.38) | 6.5 (0.37) | 7.1 (0.45) | 7.3 (0.44)
  Change at Day 8: number analyzed (Participants) | 20 | 20 | 21 | 21 | 19 | 19 | 20 | 20
  Change at Day 8 | -3.9 (0.49) | -2.0 (0.40) | -3.7 (0.53) | -2.3 (0.35) | -3.2 (0.34) | -1.9 (0.40) | -3.7 (0.46) | -2.0 (0.39)
Statistical Analysis 1: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Vehicle QD: Age Group >=12 Years; Change at Day 8, Intra-participant: Mixed effect model for repeated measures included the fixed effect of visit, and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -1.9, 95% CI 2-sided [-3.1 to -0.7], Standard Error of Mean 0.56
Statistical Analysis 2: Comparison: Crisaborole 2% BID: Age Group >=12 Years vs Vehicle BID: Age Group >=12 Years; [analysis description as in outcome 3, analysis 1]; Test type: Other; Least squares mean of difference = -1.4, 95% CI 2-sided [-2.7 to -0.2], Standard Error of Mean 0.60
Statistical Analysis 3: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Vehicle QD: Age Group 2 to 11 Years; [analysis description as in outcome 3, analysis 1]; Test type: Other; Least squares mean of difference = -1.2, 95% CI 2-sided [-2.2 to -0.2], Standard Error of Mean 0.49
Statistical Analysis 4: Comparison: Crisaborole 2% BID: Age Group 2 to 11 Years vs Vehicle BID: Age Group 2 to 11 Years; [analysis description as in outcome 3, analysis 1]; Test type: Other; Least squares mean of difference = -1.7, 95% CI 2-sided [-2.8 to -0.5], Standard Error of Mean 0.55
Statistical Analysis 5: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Crisaborole 2% BID: Age Group >=12 Years; Change at Day 8, Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen, visit, dosing regimen-by-visit interaction, and baseline value and the covariance structure UN was used; Test type: Other; Difference of least square mean = -0.1, 95% CI 2-sided [-1.5 to 1.3], Standard Error of Mean 0.69
Statistical Analysis 6: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Crisaborole 2% BID: Age Group 2 to 11 Years; [analysis description as in outcome 3, analysis 5]; Test type: Other; Difference of least square mean = -0.1, 95% CI 2-sided [-1.2 to 1.0], Standard Error of Mean 0.54

4. Secondary Outcome: Change From Baseline in Investigator's Static Global Assessment (ISGA) Score in Target Lesions at Day 8 and Day 15
Description: ISGA assessed the severity of AD on a 5-point scale ranged from 0 (clear) to 4 (severe), where higher scores indicated higher degree of AD. Grades for classification of severity: 0= clear (minor residual hypo/hyper pigmentation, no erythema or induration or papulation, no oozing or crusting), 1= almost clear (trace faint pink erythema, with barely perceptible induration or papulation and no oozing or crusting), 2= mild (faint pink erythema with mild induration or papulation and no oozing or crusting), 3= moderate (pink-red erythema with moderate induration or papulation with or without oozing or crusting) and 4= severe (deep or bright red erythema with severe induration or papulation and with oozing or crusting).
Time Frame: Baseline, Day 8, Day 15
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Crisaborole 2% QD: Age Group >=12 Years | Vehicle QD: Age Group >=12 Years | Crisaborole 2% BID: Age Group >=12 Years | Vehicle BID: Age Group >=12 Years | Crisaborole 2% QD: Age Group 2 to 11 Years | Vehicle QD: Age Group 2 to 11 Years | Crisaborole 2% BID: Age Group 2 to 11 Years | Vehicle BID: Age Group 2 to 11 Years
Number analyzed (Participants) | 20 | 20 | 21 | 21 | 20 | 20 | 20 | 20
units on a scale
  Baseline | 3.0 (0.0) | 3.0 (0.0) | 3.0 (0.0) | 3.0 (0.0) | 3.0 (0.0) | 3.0 (0.0) | 3.0 (0.0) | 3.0 (0.0)
  Change at Day 8: number analyzed (Participants) | 20 | 20 | 21 | 21 | 19 | 19 | 20 | 20
  Change at Day 8 | -1.3 (0.18) | -0.8 (0.12) | -1.1 (0.20) | -0.7 (0.12) | -1.4 (0.19) | -1.0 (0.20) | -1.2 (0.18) | -0.8 (0.16)
  Change at Day 15 | -1.9 (0.19) | -1.0 (0.15) | -1.9 (0.19) | -1.1 (0.19) | -1.8 (0.22) | -1.1 (0.19) | -1.9 (0.16) | -0.9 (0.20)
Statistical Analysis 1: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Vehicle QD: Age Group >=12 Years; [analysis description as in outcome 3, analysis 1]; Test type: Other; Least squares mean of difference = -0.5, 95% CI 2-sided [-0.9 to -0.1], Standard Error of Mean 0.17
Statistical Analysis 2: Comparison: Crisaborole 2% BID: Age Group >=12 Years vs Vehicle BID: Age Group >=12 Years; [analysis description as in outcome 3, analysis 1]; Test type: Other; Least squares mean of difference = -0.4, 95% CI 2-sided [-0.9 to 0.0], Standard Error of Mean 0.21
Statistical Analysis 3: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Vehicle QD: Age Group 2 to 11 Years; [analysis description as in outcome 3, analysis 1]; Test type: Other; Least squares mean of difference = -0.3, 95% CI 2-sided [-0.8 to 0.1], Standard Error of Mean 0.23
Statistical Analysis 4: Comparison: Crisaborole 2% BID: Age Group 2 to 11 Years vs Vehicle BID: Age Group 2 to 11 Years; [analysis description as in outcome 3, analysis 1]; Test type: Other; Least squares mean of difference = -0.4, 95% CI 2-sided [-0.8 to 0.0], Standard Error of Mean 0.20
Statistical Analysis 5: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Crisaborole 2% BID: Age Group >=12 Years; [analysis description as in outcome 3, analysis 5]; Test type: Other; Difference of least square mean = 0.1, 95% CI 2-sided [-0.4 to 0.6], Standard Error of Mean 0.27
Statistical Analysis 6: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Crisaborole 2% BID: Age Group 2 to 11 Years; [analysis description as in outcome 3, analysis 5]; Test type: Other; Difference of least square mean = 0.2, 95% CI 2-sided [-0.3 to 0.7], Standard Error of Mean 0.26
Statistical Analysis 7: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Vehicle QD: Age Group >=12 Years; [analysis description as in outcome 1, analysis 2]; Test type: Other; Least squares mean of difference = -0.9, 95% CI 2-sided [-1.4 to -0.4], Standard Error of Mean 0.22
Statistical Analysis 8: Comparison: Crisaborole 2% BID: Age Group >=12 Years vs Vehicle BID: Age Group >=12 Years; [analysis description as in outcome 1, analysis 2]; Test type: Other; Least squares mean of difference = -0.7, 95% CI 2-sided [-1.2 to -0.2], Standard Error of Mean 0.25
Statistical Analysis 9: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Vehicle QD: Age Group 2 to 11 Years; [analysis description as in outcome 1, analysis 2]; Test type: Other; Least squares mean of difference = -0.7, 95% CI 2-sided [-1.2 to -0.2], Standard Error of Mean 0.24
Statistical Analysis 10: Comparison: Crisaborole 2% BID: Age Group 2 to 11 Years vs Vehicle BID: Age Group 2 to 11 Years; [analysis description as in outcome 1, analysis 2]; Test type: Other; Least squares mean of difference = -1.0, 95% CI 2-sided [-1.4 to -0.6], Standard Error of Mean 0.21
Statistical Analysis 11: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Crisaborole 2% BID: Age Group >=12 Years; Change at Day 15, Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen, visit, dosing regimen-by-visit interaction, and baseline value and the covariance structure UN was used; Test type: Other; Difference of least square mean = 0.0, 95% CI 2-sided [-0.5 to 0.6], Standard Error of Mean 0.27
Statistical Analysis 12: Comparison: Vehicle QD: Age Group 2 to 11 Years vs Vehicle BID: Age Group 2 to 11 Years; [analysis description as in outcome 4, analysis 11]; Test type: Other; Difference of least square mean = -0.1, 95% CI 2-sided [-0.7 to 0.5], Standard Error of Mean 0.28

5. Secondary Outcome: Change From Baseline in Peak Pruritus Numerical Rating Scale (NRS) in Target Lesions up to Day 15 in Participants Aged 12 Years or More
Description: The severity of itch (pruritus) due to AD at the target lesion was assessed using the peak pruritus NRS. Participants aged 12 years or more, were asked to rate their itch severity at the worst moment during the past 24 hours on a scale ranging from 0 (no itch) to 10 (worst itch imaginable); higher scores represented more severe itch.
Time Frame: Baseline, Day 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Crisaborole 2% QD: Age Group >=12 Years | Vehicle QD: Age Group >=12 Years | Crisaborole 2% BID: Age Group >=12 Years | Vehicle BID: Age Group >=12 Years
Number analyzed (Participants) | 20 | 20 | 21 | 21
units on a scale
  Baseline | 5.3 (0.59) | 5.3 (0.57) | 5.1 (0.47) | 5.3 (0.43)
  Change at Day 2 | -1.3 (0.45) | -0.7 (0.38) | -0.6 (0.20) | -0.5 (0.37)
  Change at Day 3 | -1.7 (0.51) | -1.1 (0.49) | -1.4 (0.30) | -1.2 (0.36)
  Change at Day 4 | -2.5 (0.53) | -1.2 (0.55) | -2.0 (0.32) | -1.2 (0.44)
  Change at Day 5 | -2.6 (0.54) | -1.5 (0.46) | -2.6 (0.37) | -1.8 (0.40)
  Change at Day 6 | -2.8 (0.48) | -1.6 (0.51) | -2.2 (0.45) | -1.9 (0.46)
  Change at Day 7 | -2.9 (0.50) | -1.7 (0.56) | -2.5 (0.39) | -2.1 (0.45)
  Change at Day 8 | -3.2 (0.49) | -2.0 (0.56) | -2.8 (0.40) | -2.2 (0.48)
  Change at Day 9 | -3.2 (0.51) | -1.6 (0.55) | -2.7 (0.57) | -2.3 (0.46)
  Change at Day 10 | -3.3 (0.53) | -1.7 (0.61) | -3.0 (0.44) | -2.0 (0.58)
  Change at Day 11 | -3.5 (0.54) | -2.0 (0.55) | -3.1 (0.41) | -2.3 (0.49)
  Change at Day 12 | -3.5 (0.60) | -2.3 (0.58) | -3.3 (0.44) | -2.3 (0.50)
  Change at Day 13 | -3.4 (0.62) | -2.3 (0.57) | -3.5 (0.45) | -2.4 (0.46)
  Change at Day 14 | -3.3 (0.64) | -2.1 (0.65) | -3.6 (0.43) | -2.6 (0.47)
  Change at Day 15 | -3.5 (0.63) | -2.0 (0.63) | -3.7 (0.47) | -2.9 (0.46)
Statistical Analysis 1: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Vehicle QD: Age Group >=12 Years; Change at Day 2, Intra-participant: Mixed effect model for repeated measures included the fixed effect of day, and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -0.6, 95% CI 2-sided [-1.0 to -0.2], Standard Error of Mean 0.20
Statistical Analysis 2: Comparison: Crisaborole 2% BID: Age Group >=12 Years vs Vehicle BID: Age Group >=12 Years; [analysis description as in outcome 5, analysis 1]; Test type: Other; Least squares mean of difference = -0.1, 95% CI 2-sided [-0.7 to 0.5], Standard Error of Mean 0.28
Statistical Analysis 3: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Crisaborole 2% BID: Age Group >=12 Years; Change at Day 2, Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen, day, dosing regimen-by-day interaction, and baseline value and the covariance structure UN was used; Test type: Other; Difference of least squares mean = 0.6, 95% CI 2-sided [-0.5 to 1.7], Standard Error of Mean 0.54
Statistical Analysis 4: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Vehicle QD: Age Group >=12 Years; Change at Day 3, Intra-participant: Mixed effect model for repeated measures included the fixed effect of day, and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -0.6, 95% CI 2-sided [-1.3 to 0.1], Standard Error of Mean 0.32
Statistical Analysis 5: Comparison: Crisaborole 2% BID: Age Group >=12 Years vs Vehicle BID: Age Group >=12 Years; [analysis description as in outcome 5, analysis 4]; Test type: Other; Least squares mean of difference = -0.2, 95% CI 2-sided [-0.9 to 0.4], Standard Error of Mean 0.32
Statistical Analysis 6: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Crisaborole 2% BID: Age Group >=12 Years; Change at Day 3, Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen, day, dosing regimen-by-day interaction, and baseline value and the covariance structure UN was used; Test type: Other; Difference of least square mean = 0.2, 95% CI 2-sided [-0.9 to 1.3], Standard Error of Mean 0.55
Statistical Analysis 7: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Vehicle QD: Age Group >=12 Years; Change at Day 4, Intra-participant: Mixed effect model for repeated measures included the fixed effect of day, and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -1.3, 95% CI 2-sided [-2.1 to -0.5], Standard Error of Mean 0.38
Statistical Analysis 8: Comparison: Crisaborole 2% BID: Age Group >=12 Years vs Vehicle BID: Age Group >=12 Years; [analysis description as in outcome 5, analysis 7]; Test type: Other; Least squares mean of difference = -0.8, 95% CI 2-sided [-1.5 to -0.1], Standard Error of Mean 0.34
Statistical Analysis 9: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Crisaborole 2% BID: Age Group >=12 Years; Change at Day 4, Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen, day, dosing regimen-by-day interaction, and baseline value and the covariance structure UN was used; Test type: Other; Difference of least square mean = 0.4, 95% CI 2-sided [-0.6 to 1.4], Standard Error of Mean 0.50
Statistical Analysis 10: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Vehicle QD: Age Group >=12 Years; Change at Day 5, Intra-participant: Mixed effect model for repeated measures included the fixed effect of day, and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -1.1, 95% CI 2-sided [-1.9 to -0.3], Standard Error of Mean 0.40
Statistical Analysis 11: Comparison: Crisaborole 2% BID: Age Group >=12 Years vs Vehicle BID: Age Group >=12 Years; [analysis description as in outcome 5, analysis 10]; Test type: Other; Least squares mean of difference = -0.8, 95% CI 2-sided [-1.5 to -0.1], Standard Error of Mean 0.34
Statistical Analysis 12: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Crisaborole 2% BID: Age Group >=12 Years; Change at Day 5, Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen, day, dosing regimen-by-day interaction, and baseline value and the covariance structure UN was used; Test type: Other; Difference of least square mean = -0.1, 95% CI 2-sided [-1.1 to 1.0], Standard Error of Mean 0.52
Statistical Analysis 13: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Vehicle QD: Age Group >=12 Years; Change at Day 6, Intra-participant: Mixed effect model for repeated measures included the fixed effect of day, and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -1.3, 95% CI 2-sided [-2.1 to -0.4], Standard Error of Mean 0.42
Statistical Analysis 14: Comparison: Crisaborole 2% BID: Age Group >=12 Years vs Vehicle BID: Age Group >=12 Years; [analysis description as in outcome 5, analysis 13]; Test type: Other; Least squares mean of difference = -0.3, 95% CI 2-sided [-1.1 to 0.4], Standard Error of Mean 0.37
Statistical Analysis 15: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Crisaborole 2% BID: Age Group >=12 Years; Change at Day 6, Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen, day, dosing regimen-by-day interaction, and baseline value and the covariance structure UN was used; Test type: Other; Difference of least square mean = 0.5, 95% CI 2-sided [-0.6 to 1.5], Standard Error of Mean 0.51
Statistical Analysis 16: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Vehicle QD: Age Group >=12 Years; Change at Day 7, Intra-participant: Mixed effect model for repeated measures included the fixed effect of day, and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -1.2, 95% CI 2-sided [-2.3 to -0.1], Standard Error of Mean 0.52
Statistical Analysis 17: Comparison: Crisaborole 2% BID: Age Group >=12 Years vs Vehicle BID: Age Group >=12 Years; [analysis description as in outcome 5, analysis 16]; Test type: Other; Least squares mean of difference = -0.4, 95% CI 2-sided [-1.0 to 0.2], Standard Error of Mean 0.29
Statistical Analysis 18: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Crisaborole 2% BID: Age Group >=12 Years; Change at Day 7, Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen, day, dosing regimen-by-day interaction, and baseline value and the covariance structure UN was used; Test type: Other; Difference of least square mean = 0.3, 95% CI 2-sided [-0.6 to 1.3], Standard Error of Mean 0.45
Statistical Analysis 19: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Vehicle QD: Age Group >=12 Years; Change at Day 8, Intra-participant: Mixed effect model for repeated measures included the fixed effect of day, and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -1.2, 95% CI 2-sided [-2.0 to -0.3], Standard Error of Mean 0.40
Statistical Analysis 20: Comparison: Crisaborole 2% BID: Age Group >=12 Years vs Vehicle BID: Age Group >=12 Years; [analysis description as in outcome 5, analysis 19]; Test type: Other; Least squares mean of difference = -0.6, 95% CI 2-sided [-1.3 to 0.1], Standard Error of Mean 0.35
Statistical Analysis 21: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Crisaborole 2% BID: Age Group >=12 Years; Change at Day 8, Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen, day, dosing regimen-by-day interaction, and baseline value and the covariance structure UN was used; Test type: Other; Difference of least square mean = 0.3, 95% CI 2-sided [-0.6 to 1.2], Standard Error of Mean 0.44
Statistical Analysis 22: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Vehicle QD: Age Group >=12 Years; Change at Day 9, Intra-participant: Mixed effect model for repeated measures included the fixed effect of day, and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -1.7, 95% CI 2-sided [-2.4 to -0.9], Standard Error of Mean 0.36
Statistical Analysis 23: Comparison: Crisaborole 2% BID: Age Group >=12 Years vs Vehicle BID: Age Group >=12 Years; [analysis description as in outcome 5, analysis 22]; Test type: Other; Least squares mean of difference = -0.4, 95% CI 2-sided [-1.5 to 0.7], Standard Error of Mean 0.52
Statistical Analysis 24: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Crisaborole 2% BID: Age Group >=12 Years; Change at Day 9, Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen, day, dosing regimen-by-day interaction, and baseline value and the covariance structure UN was used; Test type: Other; Difference of least square mean = 0.5, 95% CI 2-sided [-0.7 to 1.6], Standard Error of Mean 0.59
Statistical Analysis 25: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Vehicle QD: Age Group >=12 Years; Change at Day 10, Intra-participant: Mixed effect model for repeated measures included the fixed effect of day, and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -1.6, 95% CI 2-sided [-2.3 to -0.9], Standard Error of Mean 0.31
Statistical Analysis 26: Comparison: Crisaborole 2% BID: Age Group >=12 Years vs Vehicle BID: Age Group >=12 Years; [analysis description as in outcome 5, analysis 25]; Test type: Other; Least squares mean of difference = -1.1, 95% CI 2-sided [-2.1 to -0.1], Standard Error of Mean 0.47
Statistical Analysis 27: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Crisaborole 2% BID: Age Group >=12 Years; Change at Day 10, Inter-participant: Mixed effect Model for Repeated Measures included the fixed effects of dosing regimen, day, dosing regimen-by-day interaction, and baseline value, and the covariance structure UN was used; Test type: Other; Difference of Least Squares Mean = 0.2, 95% CI 2-sided [-0.8 to 1.2], Standard Error of Mean 0.49
Statistical Analysis 28: Comparison: Crisaborole 2% BID: Age Group >=12 Years vs Vehicle BID: Age Group >=12 Years; Change at Day 11, Intra-participant: Mixed effect model for repeated measures included the fixed effect of day, and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -0.9, 95% CI 2-sided [-1.7 to 0.0], Standard Error of Mean 0.42
Statistical Analysis 29: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Vehicle QD: Age Group >=12 Years; Change at Day 11, Intra-participant: MMRM included the fixed effect of day, and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -1.5, 95% CI 2-sided [-2.3 to -0.7], Standard Error of Mean 0.38
Statistical Analysis 30: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Crisaborole 2% BID: Age Group >=12 Years; Change at Day 11, Inter-participant: Mixed effect Model for Repeated Measures included the fixed effects of dosing regimen, day, dosing regimen-by-day interaction, and baseline value, and the covariance structure UN was used; Test type: Other; Difference of Least Squares Mean = 0.2, 95% CI 2-sided [-0.7 to 1.1], Standard Error of Mean 0.44
Statistical Analysis 31: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Vehicle QD: Age Group >=12 Years; Change at Day 12, Intra-participant: Mixed effect model for repeated measures included the fixed effect of day, and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -1.3, 95% CI 2-sided [-2.0 to -0.5], Standard Error of Mean 0.34
Statistical Analysis 32: Comparison: Crisaborole 2% BID: Age Group >=12 Years vs Vehicle BID: Age Group >=12 Years; [analysis description as in outcome 5, analysis 31]; Test type: Other; Least squares mean of difference = -1.0, 95% CI 2-sided [-2.0 to 0.0], Standard Error of Mean 0.47
Statistical Analysis 33: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Crisaborole 2% BID: Age Group >=12 Years; Change at Day 12, Inter-participant: Mixed effect Model for Repeated Measures included the fixed effects of dosing regimen, day, dosing regimen-by-day interaction, and baseline value, and the covariance structure UN was used; Test type: Other; Difference of Least Squares Mean = 0.1, 95% CI 2-sided [-0.9 to 1.2], Standard Error of Mean 0.52
Statistical Analysis 34: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Vehicle QD: Age Group >=12 Years; Change at Day 13, Intra-participant: Mixed effect model for repeated measures included the fixed effect of day, and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -1.1, 95% CI 2-sided [-1.8 to -0.3], Standard Error of Mean 0.35
Statistical Analysis 35: Comparison: Crisaborole 2% BID: Age Group >=12 Years vs Vehicle BID: Age Group >=12 Years; [analysis description as in outcome 5, analysis 34]; Test type: Other; Least squares mean of difference = -1.0, 95% CI 2-sided [-2.0 to -0.1], Standard Error of Mean 0.47
Statistical Analysis 36: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Crisaborole 2% BID: Age Group >=12 Years; Change at Day 13, Inter-participant: Mixed effect Model for Repeated Measures included the fixed effects of dosing regimen, day, dosing regimen-by-day interaction, and baseline value, and the covariance structure UN was used; Test type: Other; Difference of Least Squares Mean = -0.2, 95% CI 2-sided [-1.3 to 0.9], Standard Error of Mean 0.53
Statistical Analysis 37: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Vehicle QD: Age Group >=12 Years; Change at Day 14, Intra-participant: Mixed effect model for repeated measures included the fixed effect of day, and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -1.2, 95% CI 2-sided [-1.9 to -0.5], Standard Error of Mean 0.31
Statistical Analysis 38: Comparison: Crisaborole 2% BID: Age Group >=12 Years vs Vehicle BID: Age Group >=12 Years; [analysis description as in outcome 5, analysis 37]; Test type: Other; Least squares mean of difference = -1.0, 95% CI 2-sided [-1.8 to -0.1], Standard Error of Mean 0.42
Statistical Analysis 39: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Crisaborole 2% BID: Age Group >=12 Years; Change at Day 14, Inter-participant: Mixed effect Model for Repeated Measures included the fixed effects of dosing regimen, day, dosing regimen-by-day interaction, and baseline value, and the covariance structure UN was used; Test type: Other; Difference of Least Squares Mean = -0.4, 95% CI 2-sided [-1.5 to 0.7], Standard Error of Mean 0.53
Statistical Analysis 40: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Vehicle QD: Age Group >=12 Years; Change at Day 15, Intra-participant: Mixed effect model for repeated measures included the fixed effect of day, and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -1.5, 95% CI 2-sided [-2.2 to -0.8], Standard Error of Mean 0.34
Statistical Analysis 41: Comparison: Crisaborole 2% BID: Age Group >=12 Years vs Vehicle BID: Age Group >=12 Years; [analysis description as in outcome 1, analysis 2]; Test type: Other; Least squares mean of difference = -0.8, 95% CI 2-sided [-1.5 to 0.0], Standard Error of Mean 0.36
Statistical Analysis 42: Comparison: Crisaborole 2% QD: Age Group >=12 Years vs Crisaborole 2% BID: Age Group >=12 Years; Change at Day 15, Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen, day, dosing regimen-by-day interaction, and baseline value and the covariance structure UN was used; Test type: Other; Difference of least square mean = -0.3, 95% CI 2-sided [-1.4 to 0.8], Standard Error of Mean 0.53

6. Secondary Outcome: Change From Baseline in Itch Severity Scale in Target Lesions up to Day 15 in Participants Aged Between 6 to 11 Years
Description: The itch severity scale was used for participants >=6 to 11 years of age to assess severity of itch (pruritus) due to AD at the target lesion. In this assessment, participants were asked to choose a unit that showed how itchy their skin had been on day of assessment on a 5-point scale ranging from 1= not itchy to 5= very itchy, where higher scores represented more severe itch.
Time Frame: Baseline, Day 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15
Population: Analysis population included all participants who were randomized and received greater than or equal to 1 dose of investigational product and aged between 6 to 11 years. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years: Participants in this sub-group were of age 6 to 11 Years. Investigator determined 2 target lesions of same atopic dermatitis severity in each participant at baseline (Day 1). Crisaborole ointment 2% was applied QD to 1 of the target lesions for 15 days and participants were followed up to 35 days after the end of treatment (maximum up to Day 50).
- Vehicle QD Sub-group: Age Group 6 to 11 Years: Participants in this sub-group were of age 6 to 11 Years. Investigator determined 2 target lesions of same atopic dermatitis severity in each participant at baseline (Day 1). Vehicle was applied QD to 1 of the target lesions for 15 days and participants were followed up to 35 days after the end of treatment (maximum up to Day 50).
- Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years: Participants in this sub-group were of age 6 to 11 Years. Investigator determined 2 target lesions of same atopic dermatitis severity in each participant at baseline (Day 1). Crisaborole ointment 2% was applied BID to 1 of the target lesions for 15 days and participants were followed up to 35 days after the end of treatment (maximum up to Day 50).
- Vehicle BID Sub-group: Age Group 6 to 11 Years: Participants in this sub-group were of age 6 to 11 years. Investigator determined 2 target lesions of same atopic dermatitis severity in each participant at baseline (Day 1). Vehicle was applied BID to 1 of the target lesions for 15 days and participants were followed up to 35 days after the end of treatment (maximum up to Day 50).
Arm/Group | Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years | Vehicle QD Sub-group: Age Group 6 to 11 Years | Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years | Vehicle BID Sub-group: Age Group 6 to 11 Years
Number analyzed (Participants) | 16 | 16 | 14 | 14
units on a scale
  Baseline | 1.6 (0.33) | 1.8 (0.32) | 1.9 (0.33) | 1.6 (0.34)
  Change at Day 2 | -0.7 (0.36) | -0.3 (0.35) | -0.6 (0.45) | -0.4 (0.44)
  Change at Day 3 | -0.4 (0.35) | -0.5 (0.26) | -0.9 (0.30) | -0.3 (0.46)
  Change at Day 4 | -0.4 (0.45) | -0.4 (0.32) | -0.7 (0.46) | -0.7 (0.46)
  Change at Day 5 | -0.6 (0.41) | -0.1 (0.35) | -0.7 (0.47) | -0.3 (0.30)
  Change at Day 6 | -0.8 (0.37) | -0.4 (0.34) | -0.9 (0.38) | -0.8 (0.33)
  Change at Day 7 | -0.3 (0.46) | -0.3 (0.31) | -0.9 (0.45) | -0.8 (0.43)
  Change at Day 8 | -1.1 (0.30) | -0.7 (0.36) | -1.1 (0.44) | -0.6 (0.37)
  Change at Day 9 | -0.6 (0.38) | -0.3 (0.31) | -1.4 (0.37) | -1.0 (0.26)
  Change at Day 10 | -0.8 (0.37) | -0.4 (0.34) | -1.1 (0.33) | -0.9 (0.32)
  Change at Day 11 | -1.1 (0.34) | -0.5 (0.38) | -1.1 (0.49) | -0.7 (0.32)
  Change at Day 12 | -0.8 (0.32) | 0.1 (0.40) | -1.4 (0.37) | -0.7 (0.45)
  Change at Day 13 | -0.8 (0.37) | -0.2 (0.34) | -1.4 (0.37) | -0.7 (0.44)
  Change at Day 14 | -0.9 (0.36) | -0.4 (0.31) | -1.3 (0.41) | -1.0 (0.36)
  Change at Day 15 | -0.8 (0.38) | -0.6 (0.26) | -1.3 (0.44) | -0.9 (0.38)
Statistical Analysis 1: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Vehicle QD Sub-group: Age Group 6 to 11 Years; Change at Day 2, Intra-participant: Mixed effect Model for Repeated Measures included the fixed effect of day and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -0.4, 95% CI 2-sided [-1.0 to 0.2], Standard Error of Mean 0.27
Statistical Analysis 2: Comparison: Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years vs Vehicle BID Sub-group: Age Group 6 to 11 Years; Change at Day 2, Intra-participant: Mixed effect model for repeated measures includes the fixed effect of day and the covariance structure AR1 is used; Test type: Other; Least squares mean of difference = -0.3, 95% CI 2-sided [-1.1 to 0.5], Standard Error of Mean 0.41
Statistical Analysis 3: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years; Change at Day 2, Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen day dosing regimen-by-day interaction and baseline value and the covariance structure UN was used; Test type: Other; Difference of least squares mean = 0.3, 95% CI 2-sided [-0.5 to 1.1], Standard Error of Mean 0.40
Statistical Analysis 4: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Vehicle QD Sub-group: Age Group 6 to 11 Years; Change at Day 3, Intra-participant: Mixed effect Model for Repeated Measures included the fixed effect of day and the covariance structure UN was used; Test type: Other; Least squares mean of difference = 0.1, 95% CI 2-sided [-0.6 to 0.7], Standard Error of Mean 0.30
Statistical Analysis 5: Comparison: Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years vs Vehicle BID Sub-group: Age Group 6 to 11 Years; Change at Day 3, Intra-participant: Mixed effect model for repeated measures includes the fixed effect of day and the covariance structure AR1 is used; Test type: Other; Least squares mean of difference = -0.6, 95% CI 2-sided [-1.5 to 0.2], Standard Error of Mean 0.41
Statistical Analysis 6: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years; Change at Day 3, Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen day dosing regimen-by-day interaction and baseline value and the covariance structure UN was used; Test type: Other; Difference of least squares mean = -0.2, 95% CI 2-sided [-1.0 to 0.5], Standard Error of Mean 0.36
Statistical Analysis 7: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Vehicle QD Sub-group: Age Group 6 to 11 Years; Change at Day 4, Intra-participant: Mixed effect Model for Repeated Measures included the fixed effect of day and the covariance structure UN was used; Test type: Other; Least squares mean of difference = 0.0, 96% CI 2-sided [-1.1 to 1.1], Standard Error of Mean 0.52
Statistical Analysis 8: Comparison: Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years vs Vehicle BID Sub-group: Age Group 6 to 11 Years; Change at Day 4, Intra-participant: Mixed effect model for repeated measures includes the fixed effect of day and the covariance structure AR1 is used; Test type: Other; Least squares mean of difference = 0.0, 95% CI 2-sided [-0.8 to 0.8], Standard Error of Mean 0.41
Statistical Analysis 9: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years; Change at Day 4, Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen day dosing regimen-by-day interaction and baseline value and the covariance structure UN was used; Test type: Other; Difference of least squares mean = 0.0, 95% CI 2-sided [-0.9 to 0.8], Standard Error of Mean 0.43
Statistical Analysis 10: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Vehicle QD Sub-group: Age Group 6 to 11 Years; Change at Day 5, Intra-participant: Mixed effect Model for Repeated Measures included the fixed effect of day and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -0.4, 95% CI 2-sided [-1.2 to 0.3], Standard Error of Mean 0.36
Statistical Analysis 11: Comparison: Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years vs Vehicle BID Sub-group: Age Group 6 to 11 Years; Change at Day 5, Intra-participant: Mixed effect model for repeated measures includes the fixed effect of day and the covariance structure AR1 is used; Test type: Other; Least squares mean of difference = -0.4, 95% CI 2-sided [-1.2 to 0.4], Standard Error of Mean 0.41
Statistical Analysis 12: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years; Change at Day 5, Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen day dosing regimen-by-day interaction and baseline value and the covariance structure UN was used; Test type: Other; Difference of least squares mean = 0.1, 95% CI 2-sided [-0.8 to 1.0], Standard Error of Mean 0.44
Statistical Analysis 13: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Vehicle QD Sub-group: Age Group 6 to 11 Years; Change at Day 6, Intra-participant: Mixed effect Model for Repeated Measures included the fixed effect of day and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -0.3, 95% CI 2-sided [-1.2 to 0.6], Standard Error of Mean 0.42
Statistical Analysis 14: Comparison: Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years vs Vehicle BID Sub-group: Age Group 6 to 11 Years; Change at Day 6, Intra-participant: Mixed effect model for repeated measures includes the fixed effect of day and the covariance structure AR1 is used; Test type: Other; Least squares mean of difference = -0.1, 95% CI 2-sided [-0.9 to 0.7], Standard Error of Mean 0.41
Statistical Analysis 15: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years; Change at Day 6, Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen day dosing regimen-by-day interaction and baseline value and the covariance structure UN was used; Test type: Other; Difference of least squares mean = 0.1, 95% CI 2-sided [-0.5 to 0.8], Standard Error of Mean 0.33
Statistical Analysis 16: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Vehicle QD Sub-group: Age Group 6 to 11 Years; Change at Day 7, Intra-participant: Mixed effect Model for Repeated Measures included the fixed effect of day and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -0.1, 95% CI 2-sided [-1.0 to 0.9], Standard Error of Mean 0.43
Statistical Analysis 17: Comparison: Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years vs Vehicle BID Sub-group: Age Group 6 to 11 Years; Change at Day 7, Intra-participant: Mixed effect model for repeated measures includes the fixed effect of day and the covariance structure AR1 is used; Test type: Other; Least squares mean of difference = -0.1, 95% CI 2-sided [-1.0 to 0.7], Standard Error of Mean 0.41
Statistical Analysis 18: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years; Change at Day 7, Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen day dosing regimen-by-day interaction and baseline value and the covariance structure UN was used; Test type: Other; Difference of least squares mean = -0.4, 95% CI 2-sided [-1.2 to 0.5], Standard Error of Mean 0.42
Statistical Analysis 19: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Vehicle QD Sub-group: Age Group 6 to 11 Years; Change at Day 8, Intra-participant: Mixed effect Model for Repeated Measures included the fixed effect of day and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -0.4, 95% CI 2-sided [-1.3 to 0.5], Standard Error of Mean 0.42
Statistical Analysis 20: Comparison: Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years vs Vehicle BID Sub-group: Age Group 6 to 11 Years; Change at Day 8, Intra-participant: Mixed effect model for repeated measures includes the fixed effect of day and the covariance structure AR1 is used; Test type: Other; Least squares mean of difference = -0.6, 95% CI 2-sided [-1.4 to 0.2], Standard Error of Mean 0.41
Statistical Analysis 21: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years; Change at Day 8, Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen day dosing regimen-by-day interaction and baseline value and the covariance structure UN was used; Test type: Other; Difference of least squares mean = 0.2, 95% CI 2-sided [-0.5 to 0.8], Standard Error of Mean 0.32
Statistical Analysis 22: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Vehicle QD Sub-group: Age Group 6 to 11 Years; Change at Day 9, Intra-participant: Mixed effect Model for Repeated Measures included the fixed effect of day and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -0.3, 95% CI 2-sided [-1.2 to 0.6], Standard Error of Mean 0.44
Statistical Analysis 23: Comparison: Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years vs Vehicle BID Sub-group: Age Group 6 to 11 Years; Change at Day 9, Intra-participant: Mixed effect model for repeated measures includes the fixed effect of day and the covariance structure AR1 is used; Test type: Other; Least squares mean of difference = -0.4, 95% CI 2-sided [-1.2 to 0.4], Standard Error of Mean 0.41
Statistical Analysis 24: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years; Change at Day 9, Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen day dosing regimen-by-day interaction and baseline value and the covariance structure UN was used; Test type: Other; Difference of least squares mean = -0.6, 95% CI 2-sided [-1.2 to 0.1], Standard Error of Mean 0.33
Statistical Analysis 25: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Vehicle QD Sub-group: Age Group 6 to 11 Years; Change at Day 10, Intra-participant: Mixed effect Model for Repeated Measures included the fixed effect of day and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -0.3, 95% CI 2-sided [-1.3 to 0.7], Standard Error of Mean 0.45
Statistical Analysis 26: Comparison: Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years vs Vehicle BID Sub-group: Age Group 6 to 11 Years; Change at Day 10, Intra-participant: Mixed effect model for repeated measures includes the fixed effect of day and the covariance structure AR1 is used; Test type: Other; Least squares mean of difference = -0.2, 95% CI 2-sided [-1.0 to 0.6], Standard Error of Mean 0.41
Statistical Analysis 27: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years; Change at Day 10, Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen day dosing regimen-by-day interaction and baseline value and the covariance structure UN was used; Test type: Other; Difference of least squares mean = -0.1, 95% CI 2-sided [-0.8 to 0.5], Standard Error of Mean 0.31
Statistical Analysis 28: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Vehicle QD Sub-group: Age Group 6 to 11 Years; Change at Day 11, Intra-participant: Mixed effect Model for Repeated Measures included the fixed effect of day and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -0.6, 95% CI 2-sided [-1.6 to 0.3], Standard Error of Mean 0.45
Statistical Analysis 29: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years; Change at Day 11, Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen day dosing regimen-by-day interaction and baseline value and the covariance structure UN was used; Test type: Other; Difference of least squares mean = 0.3, 95% CI 2-sided [-0.4 to 1.0], Standard Error of Mean 0.36
Statistical Analysis 30: Comparison: Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years vs Vehicle BID Sub-group: Age Group 6 to 11 Years; Change at Day 11, Intra-participant: Mixed effect model for repeated measures includes the fixed effect of day and the covariance structure AR1 is used; Test type: Other; Least squares mean of difference = -0.4, 95% CI 2-sided [-1.2 to 0.5], Standard Error of Mean 0.41
Statistical Analysis 31: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Vehicle QD Sub-group: Age Group 6 to 11 Years; Change at Day 12, Intra-participant: Mixed effect Model for Repeated Measures included the fixed effect of day and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -0.9, 95% CI 2-sided [-1.9 to 0.0], Standard Error of Mean 0.43
Statistical Analysis 32: Comparison: Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years vs Vehicle BID Sub-group: Age Group 6 to 11 Years; Change at Day 12, Intra-participant: Mixed effect model for repeated measures includes the fixed effect of day and the covariance structure AR1 is used; Test type: Other; Least squares mean of difference = -0.6, 95% CI 2-sided [-1.5 to 0.2], Standard Error of Mean 0.41
Statistical Analysis 33: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years; Change at Day 12, Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen day dosing regimen-by-day interaction and baseline value and the covariance structure UN was used; Test type: Other; Difference of least squares mean = -0.3, 95% CI 2-sided [-1.0 to 0.5], Standard Error of Mean 0.37
Statistical Analysis 34: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Vehicle QD Sub-group: Age Group 6 to 11 Years; Change at Day 13, Intra-participant: Mixed effect Model for Repeated Measures included the fixed effect of day and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -0.6, 95% CI 2-sided [-1.5 to 0.4], Standard Error of Mean 0.44
Statistical Analysis 35: Comparison: Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years vs Vehicle BID Sub-group: Age Group 6 to 11 Years; Change at Day 13, Intra-participant: Mixed effect model for repeated measures includes the fixed effect of day and the covariance structure AR1 is used; Test type: Other; Least squares mean of difference = -0.6, 95% CI 2-sided [-1.5 to 0.2], Standard Error of Mean 0.41
Statistical Analysis 36: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years; Change at Day 13, Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen day dosing regimen-by-day interaction and baseline value and the covariance structure UN was used; Test type: Other; Least squares mean = -0.4, 95% CI 2-sided [-1.1 to 0.3], Standard Error of Mean 0.34
Statistical Analysis 37: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Vehicle QD Sub-group: Age Group 6 to 11 Years; Change at Day 14, Intra-participant: Mixed effect Model for Repeated Measures included the fixed effect of day and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -0.5, 95% CI 2-sided [-1.4 to 0.4], Standard Error of Mean 0.42
Statistical Analysis 38: Comparison: Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years vs Vehicle BID Sub-group: Age Group 6 to 11 Years; Change at Day 14, Intra-participant: Mixed effect model for repeated measures includes the fixed effect of day and the covariance structure AR1 is used; Test type: Other; Least squares mean of difference = -0.3, 95% CI 2-sided [-1.1 to 0.5], Standard Error of Mean 0.41
Statistical Analysis 39: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years; Change at Day 14, Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen day dosing regimen-by-day interaction and baseline value and the covariance structure UN was used; Test type: Other; Difference of least squares mean = -0.2, 95% CI 2-sided [-1.0 to 0.6], Standard Error of Mean 0.39
Statistical Analysis 40: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Vehicle QD Sub-group: Age Group 6 to 11 Years; Change at Day 15, Intra-participant: Mixed effect Model for Repeated Measures included the fixed effect of day and the covariance structure UN was used; Test type: Other; Least squares mean of difference = -0.2, 95% CI 2-sided [-0.9 to 0.5], Standard Error of Mean 0.34
Statistical Analysis 41: Comparison: Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years vs Vehicle BID Sub-group: Age Group 6 to 11 Years; Change at Day 15, Intra-participant: Mixed effect model for repeated measures includes the fixed effect of day and the covariance structure AR1 is used; Test type: Other; Least squares mean of difference = -0.4, 95% CI 2-sided [-1.2 to 0.5], Standard Error of Mean 0.41
Statistical Analysis 42: Comparison: Crisaborole 2% QD Sub-group: Age Group 6 to 11 Years vs Crisaborole 2% BID Sub-group: Age Group 6 to 11 Years; Change at Day 15, Inter-participant: Mixed effect model for repeated measures included the fixed effects of dosing regimen day dosing regimen-by-day interaction and baseline value and the covariance structure UN was used; Test type: Other; Difference of least squares mean = -0.2, 95% CI 2-sided [-1.0 to 0.6], Standard Error of Mean 0.39

7. Secondary Outcome: Change From Baseline in Observer Reported Itch Severity Numerical Rating Scale in Target Lesions up to Day 15 in Participants Aged Between 2 to 11 Years
Description: Observer reported itch severity NRS was used for participants >=2 and < 12 years of age to assess severity of itch (pruritus) due to AD at the target lesion. Parents/caregivers (of participants) were asked to rate participants' itch (i.e. scratching, rubbing) at the worst moment during past 24 hours on a scale of 0 (no itch) to 10 (worst itch imaginable); higher scores represented more severe itch.
Time Frame: Baseline, Day 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Crisaborole 2% QD: Age Group 2 to 11 Years | Vehicle QD: Age Group 2 to 11 Years | Crisaborole 2% BID: Age Group 2 to 11 Years | Vehicle BID: Age Group 2 to 11 Years
Number analyzed (Participants) | 20 | 20 | 20 | 20
units on a scale
  Baseline | 4.7 (0.56) | 5.0 (0.50) | 5.5 (0.56) | 5.1 (0.56)
  Change at Day 2 | -0.5 (0.30) | -0.4 (0.31) | -0.7 (0.40) | -0.9 (0.50)
  Change at Day 3 | -0.7 (0.28) | -0.5 (0.35) | -1.6 (0.47) | -1.3 (0.55)
  Change at Day 4 | -0.5 (0.51) | -0.4 (0.38) | -1.8 (0.64) | -1.6 (0.58)
  Change at Day 5 | -1.4 (0.48) | -0.1 (0.60) | -2.0 (0.66) | -2.1 (0.52)
  Change at Day 6 | -1.9 (0.45) | -0.9 (0.43) | -2.7 (0.62) | -2.2 (0.66)
  Change at Day 7 | -2.0 (0.40) | -0.9 (0.45) | -3.0 (0.64) | -1.9 (0.71)
  Change at Day 8 | -2.3 (0.41) | -1.3 (0.36) | -3.3 (0.66) | -2.0 (0.70)
  Change at Day 9 | -2.0 (0.50) | -0.8 (0.42) | -3.4 (0.61) | -2.5 (0.63)
  Change at Day 10 | -2.2 (0.39) | -0.9 (0.42) | -3.9 (0.62) | -2.3 (0.65)
  Change at Day 11 | -2.4 (0.43) | -1.1 (0.45) | -3.5 (0.69) | -2.4 (0.66)
  Change at Day 12 | -2.1 (0.45) | -0.7 (0.61) | -4.1 (0.60) | -2.5 (0.65)
  Change at Day 13 | -2.1 (0.55) | -1.0 (0.50) | -4.1 (0.54) | -2.6 (0.70)
  Change at Day 14 | -2.4 (0.48) | -1.2 (0.49) | -4.3 (0.56) | -2.8 (0.66)
  Change at Day 15 | -2.5 (0.55) | -1.3 (0.45) | -4.3 (0.63) | -3.0 (0.61)
Statistical Analysis 1: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Vehicle QD: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 1]; Test type: Other; Least squares mean of difference = -0.1, 95% CI 2-sided [-0.9 to 0.7], Standard Error of Mean 0.39
Statistical Analysis 2: Comparison: Crisaborole 2% BID: Age Group 2 to 11 Years vs Vehicle BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 1]; Test type: Other; Least squares mean of difference = 0.2, 95% CI 2-sided [-0.6 to 1.0], Standard Error of Mean 0.36
Statistical Analysis 3: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Crisaborole 2% BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 3]; Test type: Other; Difference of least squares mean = 0.2, 95% CI 2-sided [-0.8 to 1.2], Standard Error of Mean 0.50
Statistical Analysis 4: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Vehicle QD: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 4]; Test type: Other; Least squares mean of difference = -0.2, 95% CI 2-sided [-0.9 to 0.5], Standard Error of Mean 0.33
Statistical Analysis 5: Comparison: Crisaborole 2% BID: Age Group 2 to 11 Years vs Vehicle BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 4]; Test type: Other; Least squares mean of difference = -0.3, 95% CI 2-sided [-1.5 to 1.0], Standard Error of Mean 0.58
Statistical Analysis 6: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Crisaborole 2% BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 6]; Test type: Other; Difference of least squares mean = -0.6, 95% CI 2-sided [-1.6 to 0.5], Standard Error of Mean 0.53
Statistical Analysis 7: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Vehicle QD: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 7]; Test type: Other; Least squares mean of difference = -0.2, 95% CI 2-sided [-1.1 to 0.8], Standard Error of Mean 0.45
Statistical Analysis 8: Comparison: Crisaborole 2% BID: Age Group 2 to 11 Years vs Vehicle BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 7]; Test type: Other; Least squares mean of difference = -0.2, 95% CI 2-sided [-1.5 to 1.1], Standard Error of Mean 0.62
Statistical Analysis 9: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Crisaborole 2% BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 9]; Test type: Other; Difference of least squares mean = -0.9, 95% CI 2-sided [-2.4 to 0.6], Standard Error of Mean 0.74
Statistical Analysis 10: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Vehicle QD: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 10]; Test type: Other; Least squares mean of difference = -1.4, 95% CI 2-sided [-2.2 to -0.5], Standard Error of Mean 0.39
Statistical Analysis 11: Comparison: Crisaborole 2% BID: Age Group 2 to 11 Years vs Vehicle BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 10]; Test type: Other; Least squares mean of difference = 0.1, 95% CI 2-sided [-1.3 to 1.5], Standard Error of Mean 0.66
Statistical Analysis 12: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Crisaborole 2% BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 12]; Test type: Other; Difference of least squares mean = -0.2, 95% CI 2-sided [-1.7 to 1.2], Standard Error of Mean 0.70
Statistical Analysis 13: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Vehicle QD: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 13]; Test type: Other; Least squares mean of difference = -1.0, 95% CI 2-sided [-2.0 to 0.0], Standard Error of Mean 0.46
Statistical Analysis 14: Comparison: Crisaborole 2% BID: Age Group 2 to 11 Years vs Vehicle BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 13]; Test type: Other; Least squares mean of difference = -0.5, 95% CI 2-sided [-1.4 to 0.5], Standard Error of Mean 0.47
Statistical Analysis 15: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Crisaborole 2% BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 15]; Test type: Other; Difference of least squares mean = -0.4, 95% CI 2-sided [-1.7 to 0.8], Standard Error of Mean 0.63
Statistical Analysis 16: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Vehicle QD: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 16]; Test type: Other; Least squares mean of difference = -1.1, 95% CI 2-sided [-2.0 to -0.2], Standard Error of Mean 0.42
Statistical Analysis 17: Comparison: Crisaborole 2% BID: Age Group 2 to 11 Years vs Vehicle BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 16]; Test type: Other; Least squares mean of difference = -1.1, 95% CI 2-sided [-2.1 to -0.1], Standard Error of Mean 0.48
Statistical Analysis 18: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Crisaborole 2% BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 18]; Test type: Other; Difference of least squares mean = -0.6, 95% CI 2-sided [-1.9 to 0.6], Standard Error of Mean 0.61
Statistical Analysis 19: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Vehicle QD: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 19]; Test type: Other; Least squares mean of difference = -1.0, 95% CI 2-sided [-2.0 to 0.0], Standard Error of Mean 0.49
Statistical Analysis 20: Comparison: Crisaborole 2% BID: Age Group 2 to 11 Years vs Vehicle BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 19]; Test type: Other; Least squares mean of difference = -1.3, 95% CI 2-sided [-2.4 to -0.2], Standard Error of Mean 0.52
Statistical Analysis 21: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Crisaborole 2% BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 21]; Test type: Other; Difference of least squares mean = -0.6, 95% CI 2-sided [-1.9 to 0.7], Standard Error of Mean 0.64
Statistical Analysis 22: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Vehicle QD: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 22]; Test type: Other; Least squares mean of difference = -1.2, 95% CI 2-sided [-2.3 to -0.1], Standard Error of Mean 0.54
Statistical Analysis 23: Comparison: Crisaborole 2% BID: Age Group 2 to 11 Years vs Vehicle BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 22]; Test type: Other; Least squares mean of difference = -0.9, 95% CI 2-sided [-1.9 to 0.1], Standard Error of Mean 0.49
Statistical Analysis 24: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Crisaborole 2% BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 24]; Test type: Other; Difference of least squares mean = -1.1, 95% CI 2-sided [-2.4 to 0.2], Standard Error of Mean 0.63
Statistical Analysis 25: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Vehicle QD: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 25]; Test type: Other; Least squares mean of difference = -1.3, 95% CI 2-sided [-2.4 to -0.1], Standard Error of Mean 0.54
Statistical Analysis 26: Comparison: Crisaborole 2% BID: Age Group 2 to 11 Years vs Vehicle BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 25]; Test type: Other; Least squares mean of difference = -1.6, 95% CI 2-sided [-2.5 to -0.7], Standard Error of Mean 0.45
Statistical Analysis 27: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Crisaborole 2% BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 27]; Test type: Other; Difference of least squares mean = -1.4, 95% CI 2-sided [-2.6 to -0.2], Standard Error of Mean 0.58
Statistical Analysis 28: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Vehicle QD: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 28]; Test type: Other; Least squares mean of difference = -1.3, 95% CI 2-sided [-2.4 to -0.1], Standard Error of Mean 0.54
Statistical Analysis 29: Comparison: Crisaborole 2% BID: Age Group 2 to 11 Years vs Vehicle BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 28]; Test type: Other; Least squares mean of difference = -1.2, 95% CI 2-sided [-2.2 to -0.1], Standard Error of Mean 0.51
Statistical Analysis 30: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Crisaborole 2% BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 29]; Test type: Other; Difference of least squares mean = -0.8, 95% CI 2-sided [-2.2 to 0.5], Standard Error of Mean 0.67
Statistical Analysis 31: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Vehicle QD: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 31]; Test type: Other; Least squares mean of difference = -1.5, 95% CI 2-sided [-2.9 to 0.0], Standard Error of Mean 0.70
Statistical Analysis 32: Comparison: Crisaborole 2% BID: Age Group 2 to 11 Years vs Vehicle BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 31]; Test type: Other; Least squares mean of difference = -1.6, 95% CI 2-sided [-2.4 to -0.7], Standard Error of Mean 0.40
Statistical Analysis 33: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Crisaborole 2% BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 33]; Test type: Other; Difference of least squares mean = -1.6, 95% CI 2-sided [-2.9 to -0.3], Standard Error of Mean 0.63
Statistical Analysis 34: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Vehicle QD: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 34]; Test type: Other; Least squares mean of difference = -1.1, 95% CI 2-sided [-2.5 to 0.3], Standard Error of Mean 0.68
Statistical Analysis 35: Comparison: Crisaborole 2% BID: Age Group 2 to 11 Years vs Vehicle BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 34]; Test type: Other; Least squares mean of difference = -1.5, 95% CI 2-sided [-2.4 to -0.6], Standard Error of Mean 0.44
Statistical Analysis 36: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Crisaborole 2% BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 36]; Test type: Other; Difference of least squares mean = -1.7, 95% CI 2-sided [-3.0 to -0.5], Standard Error of Mean 0.62
Statistical Analysis 37: Comparison: Crisaborole 2% BID: Age Group 2 to 11 Years vs Vehicle BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 37]; Test type: Other; Least squares mean of difference = -1.6, 95% CI 2-sided [-2.5 to -0.6], Standard Error of Mean 0.45
Statistical Analysis 38: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Crisaborole 2% BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 39]; Test type: Other; Difference of least squares mean = -1.6, 95% CI 2-sided [-2.8 to -0.4], Standard Error of Mean 0.59
Statistical Analysis 39: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Vehicle QD: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 37]; Test type: Other; Least squares mean of difference = -1.2, 95% CI 2-sided [-2.5 to 0.1], Standard Error of Mean 0.62
Statistical Analysis 40: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Vehicle QD: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 40]; Test type: Other; Least squares mean of difference = -1.3, 95% CI 2-sided [-2.4 to -0.1], Standard Error of Mean 0.57
Statistical Analysis 41: Comparison: Crisaborole 2% BID: Age Group 2 to 11 Years vs Vehicle BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 40]; Test type: Other; Least squares mean of difference = -1.3, 95% CI 2-sided [-2.2 to -0.3], Standard Error of Mean 0.46
Statistical Analysis 42: Comparison: Crisaborole 2% QD: Age Group 2 to 11 Years vs Crisaborole 2% BID: Age Group 2 to 11 Years; [analysis description as in outcome 6, analysis 42]; Test type: Other; Difference of least squares mean = -1.4, 95% CI 2-sided [-2.8 to -0.1], Standard Error of Mean 0.66

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) in the Target Lesions Per Medical Dictionary for Regulatory Activities (MedDRA) Preferred Term
Description: An AE was any untoward medical occurrence attributed to a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent were events between first dose of study drug and up to end of study that were absent before treatment or that worsened relative to pre-treatment state. For this outcome measure, treatment-emergent AEs occurred at each treated target lesion were summarized. MedDRA version 22.1 coding dictionary was used.
Time Frame: Day 1 up to 35 days after end of treatment (maximum up to Day 50)
Population: Safety analysis set included all participants receiving greater than or equal to 1 dose of investigational product. Treatment emergent AEs and SAEs occurred in the target lesions were planned to be summarized by treatment in each regimen for each cohort and pooled cohort.
Measure: Count of Participants; unit: Participants
Groups:
- Crisaborole 2% QD: All Age Group: Crisaborole ointment 2% was applied QD to 1 of the target lesions for 15 days and participants were followed up to 35 days after the end of treatment (maximum up to Day 50).
- Vehicle QD: All Age Group: Vehicle was applied QD to 1 of the target lesions for 15 days and participants were followed up to 35 days after the end of treatment (maximum up to Day 50).
- Crisaborole 2% BID: All Age Group: Crisaborole ointment 2% was applied BID to 1 of the target lesions for 15 days and participants were followed up to 35 days after the end of treatment (maximum up to Day 50).
- Vehicle BID: All Age Group: Vehicle was applied BID to 1 of the target lesions for 15 days and participants were followed up to 35 days after the end of treatment (maximum up to Day 50).
Arm/Group | Crisaborole 2% QD: Age Group >=12 Years | Vehicle QD: Age Group >=12 Years | Crisaborole 2% BID: Age Group >=12 Years | Vehicle BID: Age Group >=12 Years | Crisaborole 2% QD: Age Group 2 to 11 Years | Vehicle QD: Age Group 2 to 11 Years | Crisaborole 2% BID: Age Group 2 to 11 Years | Vehicle BID: Age Group 2 to 11 Years | Crisaborole 2% QD: All Age Group | Vehicle QD: All Age Group | Crisaborole 2% BID: All Age Group | Vehicle BID: All Age Group
Number analyzed (Participants) | 20 | 20 | 21 | 21 | 20 | 20 | 20 | 20 | 40 | 40 | 41 | 41
Participants
  Application site coldness | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Application site irritation | 2 | 1 | 4 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 4 | 1
  Application site pain | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0
  Application site pruritus | 2 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 2 | 2 | 1
  Application site folliculitis | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0

9. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) And Serious Adverse Events (SAEs) by Treatment Regimen
Description: An AE was any untoward medical occurrence attributed to a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; Initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to end of study that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Day 1 up to 35 days after end of treatment (maximum up to Day 50)
Population: Safety analysis set included all participants receiving greater than or equal to 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Crisaborole 2% QD + Vehicle QD, Age Group >=12 Years | Cohort 1:Crisaborole 2% BID + Vehicle BID,Age Group >=12 Years | Cohort 2:Crisaborole 2% QD + Vehicle QD, Age Group 2-11 Years | Cohort 2:Crisaborole 2% BID + Vehicle BID,Age Group 2-11 Years
Number analyzed (Participants) | 20 | 21 | 20 | 20
Participants
  Participants With AEs | 6 | 6 | 2 | 2
  Participants With SAEs | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to 35 days after end of treatment (maximum up to Day 50)
Arm/Group | Cohort 1: Crisaborole 2% QD + Vehicle QD, Age Group >=12 Years | Cohort 1:Crisaborole 2% BID + Vehicle BID,Age Group >=12 Years | Cohort 2:Crisaborole 2% QD + Vehicle QD, Age Group 2-11 Years | Cohort 2:Crisaborole 2% BID + Vehicle BID,Age Group 2-11 Years
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 6/20 | 6/21 | 2/20 | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Crisaborole 2% QD + Vehicle QD, Age Group >=12 Years (N=20) | Cohort 1:Crisaborole 2% BID + Vehicle BID,Age Group >=12 Years (N=21) | Cohort 2:Crisaborole 2% QD + Vehicle QD, Age Group 2-11 Years (N=20) | Cohort 2:Crisaborole 2% BID + Vehicle BID,Age Group 2-11 Years (N=20)
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Application site coldness (General disorders) | 0 | 1 | 0 | 0
Application site irritation (General disorders) | 3 | 4 | 0 | 0
Application site pain (General disorders) | 1 | 1 | 0 | 1
Application site pruritus (General disorders) | 3 | 2 | 0 | 1
Application site folliculitis (Infections and infestations) | 1 | 1 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT03954158/SAP_000.pdf
  • Study Protocol (2019-02-22): https://cdn.clinicaltrials.gov/large-docs/58/NCT03954158/Prot_001.pdf